CLINICAL TRIAL: NCT05442801
Title: Tropicamide Versus Cyclopentolate Objective Refraction in Pediatric Population
Brief Title: Cycloplegic Refraction Among Children
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Islamic Hospital, Jordan (Other)
Responsible Party: Principal Investigator, Hashem Abu Serhan, Principal Investigator, Islamic Hospital, Jordan
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: Cycloplegic Refraction
Record Dates: First submitted 2022-06-22; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Cycloplegia
Keywords: vision; cycloplegia; cycloplegic refraction; cyclopentolate; cyclogyl; tropicamide; mydriacil; refractive errors; latent hyperopia
MeSH Terms: conditions — Refractive Errors | interventions — Cyclopentolate; Tropicamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cyclopentolate arm (Active Comparator): To study the effect of cyclopentolate 1% for cycloplegic refractions in pediatric populations:
  Firstly, we instilled an anesthetic drop into patients' eyes. Secondly, 2 drops of cyclopentolate 1% (cyclogel) 5 minutes apart were instilled.
  Autorefraction was taken at 60 minutes after first drop instillation. Primary outcome: spherical equivalent (SE) of cycloplegic refraction at 60 minutes.
  Interventions: Drug: Cyclopentolate
- Tropicamide arm (Active Comparator): To study the effect of tropicamide 1% for cycloplegic refractions in pediatric populations:
  Firstly, we instilled an anesthetic drop into patients' eyes. Secondly, 2 drops of tropicamide 1% (mydriacil) 5 minutes apart were instilled. Autorefraction was taken at 30 minutes after first drop instillation. Primary outcome: spherical equivalent (SE) of cycloplegic refraction at 30 minutes.
  Interventions: Drug: Tropicamide

INTERVENTIONS:
Drug: Cyclopentolate — Well known eye drop used for cycloplegic refraction among children.
  Other Names: Cyclogel
  Arms: Cyclopentolate arm
Drug: Tropicamide — Well known eye drop used for cycloplegic refraction among children.
  Other Names: Mydriacil
  Arms: Tropicamide arm

SUMMARY:
The primary outcome of this study is to compare cyclopentolate 1% and tropicamide 1% for cycloplegic refractions in pediatric populations. This will be a prospective double-blinded randomized clinical trial (RCT), multi center, with randomized sequencing of cycloplegic agent; each patient received one agent at one visit, and the other agent in the next visit (2 different visits ≥ 1 week apart) within 3 months.

DETAILED DESCRIPTION:
Refractive errors assessment especially in pediatric populations is usually affected by the accommodative spasm and possibly a myopic shift in the results. Spasm of accommodation become evident as pesudomyopia or latent hyperopia. Therefore, cycloplegic refraction using cycloplegic drugs is an effective way to reduce fluctuation in accommodation or spasm of ciliary muscle. The drug of choice should have a rapid onset, appropriate cyclopegic effect and minimum side effects. Cyclopentolate and Tropicamide are well known drugs used for accommodation relaxation. Cyclopentolate is widely accepted drug of first choice for patients of all ages. Its cycloplegic effects begins at 25-75 min after administration of the drop and recovery appears through 6-24 h later.6 Ocular side effects may include irritation, lacrimation, allergic blepharoconjunctivitis, conjunctival hyperemia, and increase in intraocular pressure. Some of its systemic side effects are drowsiness, ataxia, disorientation, incoherent speech, restlessness, and visual hallucinations. Tropicamide, as an alternative, is a synthetic analog of tropic acid and is known as a safe agent for cycloplegic refraction. It characterized by a rapid onset and the cycloplegia effect appears 20-30 min after administration. Its recovery appears 6 h later with safer profile compared to cyclopentolate. Several studies have been conducted to compare the cycloplegic effect of these two agents and different results have been reported. Because of inconsistencies in the previous reported results, this randomized clinical trial was conducted to compare the cycloplegic effect between cyclopentolate and tropicamide among pediatric populations (aged between 3 and 16).

ELIGIBILITY:
Inclusion Criteria:

* Age: 3-16 years
* Brown irides; grade 4 and 5 using iris color classification system developed by Seddon et al (16)
* Duration: 2 different visits ≥ 1 weeks apart within 3 months

Exclusion Criteria:

* Abnormal red reflex (e.g., media opacity)
* History of heart or neurological diseases
* History of developmental delay
* History of a previous allergy to cycloplegic agents
* Presence of syndromes (e.g., Down's syndrome)
* History of intraocular surgery

Ages: 3 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Spherical equivalent (SE) mean difference between cyclopentolate and tropicamide | 3 months
  To study the SE of each drug and compare the mean difference between cyclopentolate and tropicamide

SECONDARY OUTCOMES:
Amplitude of accommodation | 3 months
  To measure the depth of cycloplegia mean difference between cyclopentolate and tropicamide

CONTACTS AND LOCATIONS:
Overall Officials: Wejdan Al-Thawabieh, MD, Study Director — Ophthalmology Department, Islamic Hospital, Amman, Jordan; Rami Al-Omari, MD, Study Director — Faculty of Medicine, Ophthalmology, Yarmouk University, Irbid
Locations (1):
- Islamic Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No